CLINICAL TRIAL: NCT00605761
Title: An Open Label Dose Ascending, Single Dose Study to Investigate the Pharmacokinetics of SB-656933 in Subjects With Cystic Fibrosis.
Brief Title: SD Cystic Fibrosis Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CF2110398
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung function; Anti-Inflammatory
MeSH Terms: conditions — Cystic Fibrosis | interventions — SB 656933

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cohort 1 (Experimental): 50 mg treatment
  Interventions: Drug: SB656933
- Cohort 2 (Experimental): 150 mg treatment
  Interventions: Drug: SB656933

INTERVENTIONS:
Drug: SB656933 — 50 mg treatment
  Arms: Cohort 1
Drug: SB656933 — 150 mg treatment
  Arms: Cohort 2

SUMMARY:
Subject with Cystic Fibrosis have increased clearance of many drugs. Based on pre-clinical data SB656933 was found to have low clearance and high bio-availability. This study will characterize the PK profile of a single dose of SB656933 in patients with Cystic Fibrosis. There will be two groups of subjects. The first group of subjects will receive a single dose of 50mg SB-656933. The second group of subjects will receive a single dose of up to 300 mg SB-656933. Subjects will first be screened for eligibility related to cystic fibrosis history. Safety evaluations will be undertaken and plasma samples for pharmacokinetic analysis will be collected. Additional blood samples will be taken for the pharmacodynamic endpoints CD11b and GAFS. Subjects are not required to stay overnight after their 12 hour PK sample collection on Day 1, although they may do so if they wish. On Day 2 and 3, they will return for collection of additional safety measurements, and further plasma and blood samples will be taken for 24 and 48 h pharmacokinetics and 24h CD11b/GAFS measurements, respectively.

A follow up visit (Visit 3) will be made 4-7 days after the treatment period. Subjects will be enrolled in the study for approximately 3to 7 weeks (from screening to follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Have Cystic Fibrosis
* Male greater or equal to 18 years of age or female greater or equal to 16 years of age.
* Must not be a smoker, or have smoked cigarettes or used other tobacco products regularly in the last 6 months
* Must be clinically stable with no change in symptoms or medication, no admissions to hospital, no intravenous antibiotic therapy for at least 2 weeks before study start.
* Able to perform lung function tests
* Lung test reading with FEV1 >40% predicted
* Lung test with FEV1 has not changed by >10% over past 12 months
* Must have a normal ECG.
* Women of child bearing potential must use an effective method of contraception.
* Male subjects must agree to abstain from or use a condom during sexual intercourse or use a condom/spermicide, in addition to having their female partner use another form of contraception.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal at study start.
* Signed and dated written informed consent.
* The parent/guardian must give written informed consent for the child to participate in this investigation. Adolescents must also sign the informed consent
* The subject is able to understand and follow protocol.

Exclusion Criteria:

* Any clinically abnormality found at screening that is not part of the disease of cystic fibrosis.
* any problem with pancrease
* fatty feces
* liver problems
* sudden weight loss or poor nutritional status.
* high blood pressure
* infected with the hepatitis B, hepatitis C, or HIV virus
* History of regular alcohol use
* a current non-smoker
* uses corticosteroids; regular use of high dose NSAIDs, within 2 months of study start.
* have had positive Burkholderia cepacia, or MRSA within the last 12 months
* on treatment for any mycobacterial infection
* cannot be withdrawn from oral azithromycin during study
* any marked bleeding haemoptysis in the last 12 months.
* has taken more than 4 new chemical entities within the last year.
* donate more than 500 mL within the last 56 day.
* taken part in a drug trial in 30 days or taken part in a trial with a new chemical within the last 2 months.
* on drugs that are CYP3A4, CYP2B6, CYP2C8 or OATP1B1 substrates with a narrow therapeutic index are excluded.
* using non-prescription drugs, including, herbal and dietary supplements (including St John's Wort) within 7 days or unless permitted by the Investigator and sponsor
* Consumption of grapefruit juice in last 7 seven day before study start.
* Pregnant or breast feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Blood samples | over a 48 hour time-period after single dosing with either 50mg or up tp 300mg SB656933

SECONDARY OUTCOMES:
Safety: ECG, vital signs, clinical labs | over 48hours post SB656933 dosing in both dosing sessions
Continuous adverse event monitoring | from dosing until study conclusion and follow up, 4-7 days after the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Pittsburgh, Pennsylvania